CLINICAL TRIAL: NCT01235598
Title: A 16-week Double-blind, Placebo-controlled (for Initial 2 Weeks) Randomized Period, Followed by a 24-week Open-label Extension to Assess Magnetic Resonance Image (MRI) - Verified Early Response to Certolizumab Pegol in Subjects With Active Rheumatoid Arthritis (RA)
Brief Title: Magnetic Resonance Image Verified Early Response to Certolizumab Pegol in Subjects With Active Rheumatoid Arthritis (RA)
Acronym: MARVELOUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA0028; 2009-013758-33 (EudraCT Number)
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Cimzia®; CDP870; CZP; Certolizumab Pegol; Rheumatoid Arthritis; MRI
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo followed by Certolizumab Pegol (CZP) (Other): Placebo, saline solution for sc injection at Week 0 followed by Certolizumab Pegol (CZP) 400 mg at Weeks 2, 4, and 6, then Certolizumab Pegol (CZP) 200 mg 2-weekly from Week 8 to Week 40
  Interventions: Other: Placebo; Biological: Certolizumab Pegol (CZP) 200 mg; Biological: Certolizumab Pegol (CZP) 400 mg
- Certolizumab Pegol (CZP) (Experimental): Certolizumab Pegol (CZP) 400 mg for subcutaneous injection at Weeks 0, 2 and 4 followed by 200 mg 2-weekly from Week 6 to Week 40
  Interventions: Biological: Certolizumab Pegol (CZP) 200 mg; Biological: Certolizumab Pegol (CZP) 400 mg

INTERVENTIONS:
Other: Placebo — Placebo provided for the first subcutaneous injection in single-use vials at Week 0 (2 vials required), then Certolizumab Pegol (CZP) 400 mg at Weeks 2, 4 and 6, followed by Certolizumab Pegol (CZP) 200 mg every 2 weeks from Week 8 to Week 40
  Other Names: PBO
  Arms: Placebo followed by Certolizumab Pegol (CZP)
Biological: Certolizumab Pegol (CZP) 200 mg — Placebo, saline solution for subcutaneous injection at Week 0 followed by Certolizumab Pegol (CZP) 400 mg at Weeks 2, 4, and 6, then Certolizumab Pegol (CZP) 200 mg 2-weekly from Week 8 to Week 40
  Other Names: Cimzia®; CZP; CDP870
Biological: Certolizumab Pegol (CZP) 400 mg — Placebo, saline solution for subcutaneous injection at Week 0 followed by Certolizumab Pegol (CZP) 400 mg at Weeks 2, 4, and 6, then Certolizumab Pegol (CZP) 200 mg 2-weekly from Week 8 to Week 40
  Other Names: Cimzia®; CZP; CDP870

SUMMARY:
Phase IIIb study to determine early response to Certolizumab Pegol (CZP) with Magnetic Resonance Imaging (MRI) score Outcome Measures in Rheumatoid Arthritis (RA) Clinical Trials (OMERACT) RA MRI Scoring System (RAMRIS) in subjects with RA.

DETAILED DESCRIPTION:
To identify the efficacy of Certolizumab Pegol (CZP) on synovitis in dynamic MRI parameters; to make the correlation between European League Against Rheumatism (EULAR), American College of Rheumatology (ACR)p, Disease Activity Score-28 (DAS 28) responses, and Digital XRay (DXR) assessment with reduction of synovitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of adult-onset Rheumatoid Arthritis (RA) of at least 3 months duration but no longer than 15 years
* Subjects with an active adult Rheumatoid Arthritis disease
* Subjects who have been on Disease-Modifying Anti-Rheumatic Drug (DMARD) therapy for at least 12 weeks

Exclusion Criteria:

* Subject must not have a secondary, non-inflammatory type of musculoskeletal condition (eg, osteoarthritis or fibromyalgia) that in the investigator's opinion is symptomatic enough to interfere with evaluation of the effect of study drug on the subject's primary diagnosis of Rheumatoid Arthritis (RA)
* Subject must not have a diagnosis of any other inflammatory arthritis (eg, psoriatic arthritis or ankylosing spondylitis)
* Subject must not have a history of an infected joint prosthesis at any time with prosthesis still in situ
* Subject must not have received more than 1 biological agent
* Subject must not have a history of lymphoproliferative disorder including lymphoma or signs and symptoms suggestive of lymphoproliferative disease at any time
* Subject with known Tuberculosis (TB) disease, high risk of acquiring TB infection or latent TB infection
* Subject must not have a known hypersensitivity to any components of the investigational medicinal product
* Subject must not have contraindications for Magnetic Resonance Image (MRI) and contrast agent
* Subject must not have any other condition which, in the investigator's judgement, would make them unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (10):
- Denmark (4):
  - 003, Frederiksberg
  - 002, Hellerup
  - 001, Hvidovre
  - 016, Slagelse
- Netherlands (2):
  - 012, Nijmegen
  - 010, Utrecht
- Poland (2):
  - 018, Warsaw
  - 019, Warsaw
- Sweden (2):
  - 008, Gothenburg
  - 004, Malmo

REFERENCES:
- [Derived] Ostergaard M, Jacobsson LT, Schaufelberger C, Hansen MS, Bijlsma JW, Dudek A, Rell-Bakalarska M, Staelens F, Haake R, Sundman-Engberg B, Bliddal H. MRI assessment of early response to certolizumab pegol in rheumatoid arthritis: a randomised, double-blind, placebo-controlled phase IIIb study applying MRI at weeks 0, 1, 2, 4, 8 and 16. Ann Rheum Dis. 2015 Jun;74(6):1156-63. doi: 10.1136/annrheumdis-2014-206359. Epub 2014 Dec 15. PMID 25512675
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Participant Flow refers to the Randomized Set (RS) population which consists of all subjects randomized into the study.
Pre-assignment Details: The study population consists of subjects with a diagnosis of adult-onset Rheumatoid Arthritis of at least 3 months duration but not longer than 15 years. In addition, subjects must be on Disease Modifying Anti-Rheumatic Drugs (DMARD) therapy for at least 12 weeks with a stable dose / route of administration for at least 8 weeks prior to Baseline.
Groups:
- Placebo Followed by Certolizumab Pegol (CZP): Placebo, saline solution for subcutaneous injection at Week 0 followed by Certolizumab Pegol (CZP) 400 mg at Weeks 2, 4, and 6, then Certolizumab Pegol (CZP) 200 mg 2-weekly from Week 8 to Week 40
Period: Overall Study
Arm/Group | Placebo Followed by Certolizumab Pegol (CZP) | Certolizumab Pegol (CZP)
Started | 13 | 28 (One subject was randomized to the CZP Arm but never received an injection (due to pre-treatment AE))
Completed | 12 | 24
Not Completed | 1 | 4
Not completed — Adverse Event | 0 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline characteristics refer to the Safety Set (SS) population. The Safety Population includes all subjects enrolled who received at least 1 injection of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Followed by Certolizumab Pegol (CZP) | Certolizumab Pegol (CZP) | Total
Number analyzed (Participants) | 13 | 27 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 21 | 32
  >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (14.4) | 51.3 (12.6) | 50.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 22 | 32
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Poland | 2 | 7 | 9
  Denmark | 6 | 11 | 17
  Netherlands | 1 | 3 | 4
  Sweden | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Synovitis Measured by Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) Rheumatoid Arthritis Magnetic Resonance Image Scoring System (RAMRIS) Score at Week 16 Compared to Baseline for Certolizumab Pegol Arm
Description: Rheumatoid Arthritis Magnetic Resonance Image Scoring System (RAMRIS):
  Synovitis is defined as an area in the synovial compartment that shows above normal postgadolinium enhancement of a thickness greater than the width of the normal synovium. T1-weighted images were acquired before and after the administration of intravenous contrast agent containing gadolinium. Intravenous contrast was required to demonstrate enhancing synovitis. Synovitis was scored 0 to 3 in 3 wrist regions and in each of the second through fifth metacarpophalangeal (MCP) joints. A score of 0 is normal, with no enhancement or enhancement up to the thickness of normal synovium, while scores of 1 to 3 (mild, moderate, severe) refer to increments of one-third of the presumed maximum volume of enhancing tissue in the synovial compartment. Total synovitis score ranges from a minimum of 0 to a maximum of 21. A negative value in synovitis change from Baseline score indicates an improvement.
Time Frame: From Baseline to Week 16
Population: The Analysis Population refers to the Full Analysis Set (FAS) (last observation carried forward) which consists of all randomized subjects that received at least one dose of study medication. As pre-specified in the protocol, this analysis is restricted to the Certolizumab Pegol (CZP) arm.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 27
scores on a scale | -1.0 (2.3) [-3.0 to 0]
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); A fixed-sequence stepwise hypothesis testing procedure was followed using a pre-specified set of ordered hypotheses. Hypotheses were ordered and tested in that order, beginning with change from Baseline at Week 16, and continuing to earlier time points (Week 8, 4, 2, 1 in that order) only if the previous null hypothesis of zero difference was rejected (p <0.05). Hypothesis testing was stopped if and when a non-significant result was obtained; Test type: Superiority or Other; p = 0.049, Permutation test with general scores — Two-sided p-value is presented, with p < 0.05 as the threshold for statistical significance; Median difference within group changes = -1.5, 95% CI 2-sided [-3.0 to 0.0] — Hodges-Lehmann estimate of median difference and associated exact 95 % 2-sided confidence interval are provided

2. Primary Outcome: Change in Synovitis Measured by Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) Rheumatoid Arthritis Magnetic Resonance Image Scoring System (RAMRIS) Score at Week 8 Compared to Baseline for Certolizumab Pegol Arm
Description: as for outcome 1
Time Frame: From Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 27
scores on a scale | -0.7 (2.6)
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); A fixed-sequence stepwise hypothesis testing procedure was followed using a pre-specified set of ordered hypotheses. Hypotheses were ordered and tested in that order, beginning with change from Baseline at Week 16, and continuing to earlier time points (Week 8, 4, 2, 1 in that order) only if the previous null hypothesis of zero difference was rejected (p < 0.05). Hypothesis testing was stopped if and when a non-significant result was obtained. Testing was stopped in the next step; Test type: Superiority or Other; p = 0.206, Permutation test with general scores — Two-sided p-value is presented, with p < 0.05 as the threshold for statistical significance. A fixed-sequence stepwise hypothesis testing procedure was followed using a pre-specified set of ordered hypotheses; Median Difference within group changes = -1.0, 95% CI 2-sided [-3.0 to 1.0] — Hodges-Lehmann estimate of median difference and associated exact 95 % 2-sided confidence interval are provided

3. Primary Outcome: Change in Synovitis Measured by Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) Rheumatoid Arthritis Magnetic Resonance Image Scoring System (RAMRIS) Score at Week 4 Compared to Baseline for Certolizumab Pegol Arm
Description: as for outcome 1
Time Frame: From Baseline to Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 27
scores on a scale | -0.4 (1.6)

4. Primary Outcome: Change in Synovitis Measured by Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) Rheumatoid Arthritis Magnetic Resonance Image Scoring System (RAMRIS) Score at Week 2 Compared to Baseline for Certolizumab Pegol Arm
Description: as for outcome 1
Time Frame: From Baseline to Week 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 27
scores on a scale | -0.4 (1.6)

5. Primary Outcome: Change in Synovitis Measured by Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) Rheumatoid Arthritis Magnetic Resonance Image Scoring System (RAMRIS) Score at Week 1 Compared to Baseline for Certolizumab Pegol Arm
Description: as for outcome 1
Time Frame: From Baseline to Week 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 27
scores on a scale | -0.6 (1.8)

6. Secondary Outcome: Change From Baseline to Week 16 in the Dynamic Magnetic Resonance Image (MRI) Parameter, Initiation Rate of Enhancement (IRE)
Description: Contrast enhancement can be quantified in terms of the dynamic MRI parameters initial rate of enhancement (IRE), maximum enhancement (ME), and number of voxels (Nvox) with Plateau and Washout pattern. These parameters are extracted by examining individual signal intensity versus time curves derived from defined regions of interest.
  Nvox indicates the number of voxels showing enhancement patterns. It is representative of the size or volume of enhancement and representative of underlying inflammation. The higher the value, the higher the volume .
  ME and IRE values quantify the intensity of signal within the enhancing voxels. The absolute values and changes from Baseline in the MRI parameters of IRE, ME, and Nvox of the selected hand and wrist were estimated at Weeks 1, 2, 4, 8, and 16.
  The values presented are for Proximal Interphalangeal (PIP) and Metacarpophalangeal (MCP) joints combined. A negative value in IRE change from Baseline score indicates an improvement.
Time Frame: From Baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent per second
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 22
percent per second | -0.0044 (0.0140)
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.164, Permutation test with general scores — Two-sided p-value is presented, with p <0.05 as the threshold for statistical significance. A fixed-sequence stepwise hypothesis testing procedure was followed using a pre-specified set of ordered hypotheses; Median difference within group changes = -0.0035, 95% CI 2-sided [-0.0120 to 0.0025] — Hodges-Lehmann estimate of median difference and associated exact 95 % 2-sided confidence interval are provided

7. Secondary Outcome: Change From Baseline to Week 16 in the Dynamic Magnetic Resonance Image (MRI) Parameter, Maximal Enhancement (ME)
Description: Contrast enhancement can be quantified in terms of the dynamic MRI parameters initial rate of enhancement (IRE), maximum enhancement (ME), and number of voxels (Nvox) with Plateau and Washout pattern. These parameters are extracted by examining individual signal intensity versus time curves derived from defined regions of interest.
  Nvox indicates the number of voxels showing enhancement patterns. It is representative of the size or volume of enhancement and representative of underlying inflammation. The higher the value, the higher the volume .
  ME and IRE values quantify the intensity of signal within the enhancing voxels. The absolute values and changes from Baseline in the MRI parameters of IRE, ME, and Nvox of the selected hand and wrist were estimated at Weeks 1, 2, 4, 8, and 16.
  The values presented are for Proximal Interphalangeal (PIP) and Metacarpophalangeal (MCP) joints combined. A negative value in ME change from Baseline score indicates an improvement.
Time Frame: From Baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change over pre-contrast
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 22
percent change over pre-contrast | -0.0172 (0.4459)
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.865, Permutation test with general scores — [p-value comment as in outcome 6, analysis 1]; Median difference within group changes = -0.0690, 95% CI 2-sided [-0.2010 to 0.1380] — Hodges-Lehmann estimate of median difference and associated exact 95 % 2-sided confidence interval are provided

8. Secondary Outcome: Change From Baseline to Week 16 in the Dynamic Magnetic Resonance Image (MRI) Parameter, Number of Voxels (Nvox) With Plateau and Washout Pattern
Description: Contrast enhancement can be quantified in terms of the dynamic MRI parameters initial rate of enhancement (IRE), maximum enhancement (ME), and number of voxels (Nvox) with Plateau and Washout pattern. These parameters are extracted by examining individual signal intensity versus time curves derived from defined regions of interest.
  Nvox indicates the number of voxels showing enhancement patterns. It is representative of the size or volume of enhancement and representative of underlying inflammation. The higher the value, the higher the volume .
  ME and IRE values quantify the intensity of signal within the enhancing voxels. The absolute values and changes from Baseline in the MRI parameters of IRE, ME, and Nvox of the selected hand and wrist were estimated at Weeks 1, 2, 4, 8, and 16.
  The values presented are for Proximal Interphalangeal (PIP) and Metacarpophalangeal (MCP) joints combined. A negative value in Nvox change from Baseline score indicates an improvement.
Time Frame: From Baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: voxels
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 22
voxels | -813.3 (1457.3)
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.015, Permutation test with general scores — [p-value comment as in outcome 6, analysis 1]; Median difference within group changes = -421.5, 95% CI 2-sided [-1542.5 to -47.0] — Hodges-Lehmann estimate of median difference and associated exact 95 % 2-sided confidence interval are provided

9. Secondary Outcome: Percentage of Subjects Achieving a Good European League Against Rheumatism (EULAR) Response at Week 16
Description: EULAR (European League Against Rheumatism) response: EULAR response is based upon current Disease Activity Score 28 (DAS28) level and corresponding change from Baseline in DAS28.
  Good EULAR response is defined as: DAS28 C-Reactive Protein (CRP) ≤ 3.2 and decrease from Baseline by > 1.2; moderate response is defined as achievement of one of the following:
  * DAS28(CRP) ≤ 3.2 and decrease from Baseline > 0.6 and ≤ 1.2
  * DAS28(CRP) > 3.2 and ≤ 5.1 and decrease from Baseline > 0.6
  * DAS28(CRP) > 5.1 and decrease from Baseline > 1.2
Time Frame: From Baseline to Week 16
Population: The Analysis Population refers to the Full Analysis Set (FAS) (observed case) which consists of all randomized subjects that received at least one dose of study medication.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 21 | 12
percentage of subjects
  Good Response | 71.4 | 66.7
  Moderate Response | 23.8 | 25.0
  No Response | 4.8 | 8.3

10. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Criteria (ACR20) at Week 16
Description: Subjects who meet the ACR20 criteria are those subjects with at least 20 % improvement from Baseline for Tender Joint Count (TJC), Swollen Joint Count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-Reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS).
Time Frame: From Baseline to Week 16
Population: as for outcome 9
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 22 | 12
percentage of subjects
  Response | 86.4 | 75.0
  No Response | 13.6 | 25.0

11. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Criteria (ACR50) at Week 16
Description: Subjects who meet the ACR50 criteria are those subjects with at least 50 % improvement from Baseline for Tender Joint Count (TJC), Swollen Joint Count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-Reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS).
Time Frame: From Baseline to Week 16
Population: as for outcome 9
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 22 | 12
percentage of subjects
  Response | 68.2 | 58.3
  No Response | 31.8 | 41.7

12. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Criteria (ACR70) at Week 16
Description: Subjects who meet the ACR70 criteria are those subjects with at least 70 % improvement from Baseline for Tender Joint Count (TJC), Swollen Joint Count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-Reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS).
Time Frame: From Baseline to Week 16
Population: as for outcome 9
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 22 | 12
percentage of subjects
  Response | 45.5 | 58.3
  No Response | 54.5 | 41.7

13. Secondary Outcome: Change From Baseline to Week 16 in the Disease Activity Score-28 (C-Reactive Protein) (DAS28 (CRP)) Response
Description: DAS28[CRP] is a composite index and is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) C-reactive protein (CRP in mg/l), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.36 x lognat (CRP+1) + 0.014 x Global Assessment of Arthritis + 0.96 where 28 joints are examined and a lower score indicates less disease activity. A DAS(28) score of higher than 5.1 is indicative of high disease activity whereas a DAS score below 3.2 indicates low disease activity. A patient is considered to be in remission if they have a DAS28 lower than 2.6. A negative value in DAS28[CRP] change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline to Week 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 21 | 12
units on a scale | -2.27 (0.86) | -2.50 (1.23)

14. Secondary Outcome: Percentage of Subjects Achieving Disease Activity Score 28 (DAS28 (CRP)) Remission Status (DAS28 (CRP) < 2.6) at Week 16
Description: DAS28[CRP] is a composite index and is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) C-reactive protein (CRP in mg/l), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.36 x lognat (CRP+1) + 0.014 x Global Assessment of Arthritis + 0.96 where 28 joints are examined and a lower score indicates less disease activity. A DAS(28) score of higher than 5.1 is indicative of high disease activity whereas a DAS score below 3.2 indicates low disease activity. A patient is considered to be in remission if they have a DAS28 lower than 2.6.
Time Frame: From Baseline to Week 16
Population: The Analysis Population refers to the Full Analysis Set (FAS) (observed case) which consists of all randomized subjects that received at least one dose of study medication, and had a valid Baseline efficacy assessment and at least one valid post-Baseline efficacy assessment.
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 21 | 12
percentage of subjects
  Remission | 57.1 | 58.3
  No Remission | 42.9 | 41.7

15. Secondary Outcome: Change From Baseline to Week 16 in Bone Mineral Density as Measured by Digital XRay (DXR)
Description: Radiographic assessment of bone mineral density in one hand and wrist were conducted by Digital X Ray (DXR) using a standardized imaging methodology. The hand and wrist to be assessed by DXR were the same as for the Magnetic Resonance Images (MRIs). The same hand and wrist were used for all x rays. The evaluation of all DXRs was performed centrally.
  A positive value in Bone Mineral Density change from Baseline indicates an improvement.
Time Frame: From Baseline to Week 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 20 | 11
g/cm^2 | -0.00606 (0.01185) | -0.00630 (0.01032)

16. Secondary Outcome: Change From Baseline to Week 16 in Tender Joint Count (TJC)
Description: The joint assessment was carried out on 28 joints. Swelling and tenderness were graded on a 2-point scale (answered with Yes/No). "No" indicated "Not tender"; "Yes" indicated a positive tenderness response that was defined as a positive response to questioning (tender), spontaneous response elicited (tender and winced) or withdrawal by subject on examination (tender, winced, and withdrew)." If there were missing observations in the TJC, then the remaining observations were assessed and weighted by dividing by the number of non-missing joint counts and multiplying by 28. TJC ranges from 0 to 28 with 0 indicating no tender joints and 28 indicating tenderness in all joints. A negative value in TJC change from Baseline indicates an improvement.
Time Frame: From Baseline to Week 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 23 | 12
units on a scale | -9.28 (5.85) | -9.92 (8.55)

17. Secondary Outcome: Change From Baseline to Week 16 in Swollen Joint Count (SJC)
Description: The joint assessment was carried out on 28 joints. Swelling and tenderness were graded on a 2-point scale (answered with Yes/No). "No" indicated "None" swelling response and "Yes" indicated that there was "a detectable synovial thickening with or without loss of bony contours, or bulging synovial proliferation with or without cystic characteristics." If there were missing observations in the SJC, then the remaining observations were assessed and weighted by dividing by the number of non-missing joint counts and multiplying by 28. SJC ranges from 0 to 28 with 0 indicating no swollen joints and 28 indicating swelling in all joints. A negative value in SJC change from Baseline indicates an improvement.
Time Frame: From Baseline to Week 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 23 | 12
units on a scale | -7.06 (4.67) | -7.92 (5.81)

18. Secondary Outcome: Change From Baseline to Week 16 in Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI) is a subject reported questionnaire that provides an assessment of the impact of the disease and its treatment on physical function. The HAQ-DI assesses the degree of difficulty experienced in 8 domains of daily living activities using 20 questions. The domains are dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities, and each domain (activity) consists of 2 or 3 items. For each question the level of difficulty is scored from 0 to 3 where 0 = no difficulty, 1 = some difficulty, 2 = much difficulty and 3 = unable to do. A total score is computed from the item scores using the scoring rules provided by the author (Fries, 1980). The total score ranges from 0 to 3 with lower scores meaning lower disability. A negative value in HAQ-DI change from Baseline indicates an improvement.
Time Frame: From Baseline to Week 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 23 | 12
scores on a scale | -0.54 (0.49) | -0.79 (0.49)

19. Secondary Outcome: C-Reactive Protein (CRP) Ratio to Baseline at Week 16
Description: The C-Reactive Protein (CRP) is considered a marker of inflammation in subjects with Rheumatoid Arthritis.
  A ratio to Baseline < 1 indicates an improvement.
Time Frame: From Baseline to Week 16
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Certolizumab Pegol (CZP) | Placebo Followed by Certolizumab Pegol (CZP)
Number analyzed (Participants) | 21 | 12
ratio | 0.491 (175.1) [0.179 to 0.947] | 0.219 (147.9)

20. Secondary Outcome: Correlation of Change in Synovitis From Baseline as Measured by Magnetic Resonance Image (MRI) With European League Against Rheumatism (EULAR) Response at Week 16
Description: EULAR (European League Against Rheumatism) response: EULAR response is based upon current Disease Activity Score 28 (DAS28) level and corresponding change from Baseline in DAS28.
  Good EULAR response is defined as: DAS28 C-Reactive Protein (CRP) ≤ 3.2 and decrease from Baseline by > 1.2; moderate response is defined as achievement of one of the following:
  * DAS28(CRP) ≤ 3.2 and decrease from Baseline > 0.6 and ≤ 1.2
  * DAS28(CRP) > 3.2 and ≤ 5.1 and decrease from Baseline > 0.6
  * DAS28(CRP) > 5.1 and decrease from Baseline > 1.2
  A negative correlation coefficient indicates that reductions in synovitis from Baseline to Week 16 are associated with better EULAR responses.
Time Frame: From Baseline to Week 16
Population: The Analysis Population refers to the Full Analysis Set (FAS) (observed case) which consists of all randomized subjects that received at least one dose of study medication. Correlations between the change from Baseline in total synovitis score at Week 16 and the clinical efficacy variables are restricted to the Certolizumab Pegol (CZP) arm only.
Measure: Number; unit: Spearman rank correlation coefficient
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 20
Spearman rank correlation coefficient | -0.20
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); Test type: Superiority or Other; p = 0.394, Spearman rank correlation

21. Secondary Outcome: Correlation of Change in Synovitis From Baseline as Measured by Magnetic Resonance Image (MRI) With American College of Rheumatology 20 % Criteria (ACR20) at Week 16
Description: Subjects who meet the ACR20 criteria are those subjects with at least 20 % improvement from Baseline for Tender Joint Count (TJC), Swollen Joint Count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-Reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS).
  A negative correlation coefficient indicates that reductions in synovitis from Baseline to Week 16 are associated with an ACR20 response at Week 16.
Time Frame: From Baseline to Week 16
Population: as for outcome 20
Measure: Number; unit: Spearman rank correlation coefficient
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 21
Spearman rank correlation coefficient | -0.11
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); Test type: Superiority or Other; p = 0.625, Spearman rank correlation

22. Secondary Outcome: Correlation of Change in Synovitis From Baseline as Measured by Magnetic Resonance Image (MRI) With American College of Rheumatology 50 % Criteria (ACR50) at Week 16
Description: Subjects who meet the ACR50 criteria are those subjects with at least 50 % improvement from Baseline for Tender Joint Count (TJC), Swollen Joint Count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-Reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS).
  A negative correlation coefficient indicates that reductions in synovitis from Baseline to Week 16 are associated with an ACR50 response at Week 16.
Time Frame: From Baseline to Week 16
Population: as for outcome 20
Measure: Number; unit: Spearman rank correlation coefficient
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 21
Spearman rank correlation coefficient | -0.34
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); Test type: Superiority or Other; p = 0.128, Spearman rank correlation

23. Secondary Outcome: Correlation of Change in Synovitis From Baseline as Measured by Magnetic Resonance Image (MRI) With American College of Rheumatology 70 % Criteria (ACR70) at Week 16
Description: Subjects who meet the ACR70 criteria are those subjects with at least 70 % improvement from Baseline for Tender Joint Count (TJC), Swollen Joint Count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-Reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS), 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale (PtGADA-VAS), 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale (PhGA-VAS).
  A negative correlation coefficient indicates that reductions in synovitis from Baseline to Week 16 are associated with an ACR70 response at Week 16.
Time Frame: From Baseline to Week 16
Population: as for outcome 20
Measure: Number; unit: Spearman rank correlation coefficient
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 21
Spearman rank correlation coefficient | -0.08
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); Test type: Superiority or Other; p = 0.732, Spearman rank correlation

24. Secondary Outcome: Correlation of Change in Synovitis From Baseline as Measured by Magnetic Resonance Image (MRI) With Disease Activity Score-28 (DAS28 (CRP)) Response at Week 16
Description: The DAS28(CRP) was calculated using the tender joint count (TJC) and swollen joint count (SJC), C-Reactive Protein (CRP in mg/L) and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm).
  A positive correlation coefficient indicates that reductions in synovitis from Baseline to Week 16 are associated with reductions in DAS28(CRP) at Week 16.
Time Frame: From Baseline to Week 16
Population: as for outcome 20
Measure: Number; unit: Spearman rank correlation coefficient
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 20
Spearman rank correlation coefficient | 0.19
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); Test type: Superiority or Other; p = 0.411, Spearman rank correlation

25. Secondary Outcome: Correlation of Change in Synovitis From Baseline as Measured by Magnetic Resonance Image (MRI) With Changes in Hand Bone Mineral Density as Measured by Digital XRay (DXR) at Week 16
Description: Radiographic assessment of bone mineral density in one hand and wrist were conducted by Digital X Ray (DXR) using a standardized imaging methodology. The hand and wrist to be assessed by DXR were the same as for the Magnetic Resonance Images (MRIs). The same hand and wrist were used for all x rays. The evaluation of all DXRs was performed centrally.
  A negative correlation coefficient indicates that reductions in synovitis from Baseline to Week 16 are associated with increases in bone mineral density at Week 16.
Time Frame: From Baseline to Week 16
Population: as for outcome 20
Measure: Number; unit: Spearman rank correlation coefficient
Arm/Group | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 17
Spearman rank correlation coefficient | 0.32
Statistical Analysis 1: Comparison: Certolizumab Pegol (CZP); Test type: Superiority or Other; p = 0.208, Spearman rank correlation

26. Secondary Outcome: Change From Baseline for the Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) Rheumatoid Arthritis Magnetic Resonance Image Scoring System (RAMRIS) Synovitis Score at Week 1 Placebo (PBO) Versus Certolizumab Pegol (CZP)
Description: Rheumatoid Arthritis Magnetic Resonance Image Scoring System (RAMRIS):
  Synovitis is defined as an area in the synovial compartment that shows above normal postgadolinium enhancement of a thickness greater than the width of the normal synovium. T1-weighted images were acquired before and after the administration of intravenous contrast agent containing gadolinium. Intravenous contrast was required to demonstrate enhancing synovitis. Synovitis was scored 0 to 3 in 3 wrist regions (the distal radioulnar; the radiocarpal joint; the intercarpal and carpometacarpal joints) and in each of the second through fifth metacarpophalangeal (MCP) joints. A score of 0 is normal, with no enhancement or enhancement up to the thickness of normal synovium, while scores of 1 to 3 (mild, moderate, severe) refer to increments of one-third of the presumed maximum volume of enhancing tissue in the synovial compartment.
  A negative value in synovitis change from Baseline score indicates an improvement.
Time Frame: From Baseline to Week 1
Population: The Analysis Population refers to the Full Analysis Set (FAS) (last observation carried forward) which consists of all randomized subjects that received at least one dose of study medication, and had a valid Baseline efficacy assessment and at least one valid post-Baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo Followed by Certolizumab Pegol (CZP) | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 13 | 27
scores on a scale | 0.1 (1.0) | -0.6 (1.8)
Statistical Analysis 1: Comparison: Placebo Followed by Certolizumab Pegol (CZP) vs Certolizumab Pegol (CZP); Test type: Superiority or Other; p = 0.254, Wilcoxon Rank-Sum Test — Two-sided p-value is presented, with p <0.05 as the threshold for statistical significance; Median Difference (Net) = 0.0, 95% CI 2-sided [-1.0 to 0.0] — Hodges-Lehmann estimate of median difference and associated exact 95 % 2-sided confidence interval are provided

27. Secondary Outcome: Change From Baseline for the Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) Rheumatoid Arthritis Magnetic Resonance Image Scoring System (RAMRIS) Synovitis Score at Week 2 Placebo (PBO) Versus Certolizumab Pegol (CZP)
Description: as for outcome 26
Time Frame: From Baseline to Week 2
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo Followed by Certolizumab Pegol (CZP) | Certolizumab Pegol (CZP)
Number analyzed (Participants) | 13 | 27
scores on a scale | 0.2 (1.4) | -0.4 (1.6)
Statistical Analysis 1: Comparison: Placebo Followed by Certolizumab Pegol (CZP) vs Certolizumab Pegol (CZP); Test type: Superiority or Other; p = 0.472, Wilcoxon Rank-Sum Test — Two-sided p-value is presented, with p <0.05 as the threshold for statistical significance; Median Difference (Net) = 0.0, 95% CI 2-sided [-2.0 to 1.0] — Hodges-Lehmann estimate of median difference and associated exact 95 % 2-sided confidence interval are provided

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) were reported from Baseline (Week 0) to the end of the study (Week 50).
Description: Subjects that did not receive at least one dose of Certolizumab Pegol (CZP) were excluded. Only Treatment Emergent Adverse Events (TEAEs) occurring while receiving CZP are reported.
Groups:
- Certolizumab Pegol (CZP) at Any Time: Eligible subjects were allocated to the following study treatments in a 2:1 ratio:
  * Certolizumab Pegol (CZP) 400mg for subcutaneous injection (sc) at Weeks 0, 2, and 4, followed by CZP 200mg sc and placebo (saline solution) at Week 6 and CZP 200mg at Weeks 8, 10, 12, 14, and 16 or
  * Placebo (saline solution) at Day 0 and then CZP 400mg sc at Weeks 2, 4, and 6 followed by CZP 200mg sc at Weeks 8, 10, 12, 14, and 16
Arm/Group | Certolizumab Pegol (CZP) at Any Time
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 26/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (CZP) at Any Time (N=40)
Splinter haemorrhages (Cardiac disorders) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sensory Loss (Nervous system disorders) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (CZP) at Any Time (N=40)
Nausea (Gastrointestinal disorders) | 2 (2)
Injection site pain (General disorders) | 3 (5)
Injection site discolouration (General disorders) | 2 (5)
Nodule (General disorders) | 2 (5)
Injection site swelling (General disorders) | 2 (3)
Fatigue (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (8)
Urinary tract infection (Infections and infestations) | 5 (5)
Oral herpes (Infections and infestations) | 4 (9)
Viral infection (Infections and infestations) | 4 (5)
Influenza (Infections and infestations) | 3 (3)
Pharyngitis bacterial (Infections and infestations) | 2 (5)
Abscess (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Hepatic enzyme increased (Investigations) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (3)
Tendon pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (14)
Dizziness (Nervous system disorders) | 3 (4)
Paraesthesia (Nervous system disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
Hot flush (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days